CLINICAL TRIAL: NCT00483730
Title: A Multi-centre, Double-blind, Placebo-controlled, Randomised, Parallel Group Clinical Trial to Evaluate Efficacy and Safety of Actovegin® in Diabetic Type 2 Patients With Symptomatic Diabetic Peripheral Polyneuropathy
Brief Title: Actovegin® Versus Placebo in Patients With Diabetic Polyneuropathy (AV-007-IM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Nycomed
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AV-007-IM
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Symptomatic Diabetic Peripheral Polyneuropathy
MeSH Terms: interventions — Actovegin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Deproteinised hemoderivative of calf blood (Actovegin) — Symptomatic diabetic peripheral polyneuropathy

SUMMARY:
To assess clinical efficacy and safety of Actovegin in type 2 diabetic patients with symptomatic diabetic peripheral polyneuropathy after 250 ml i.v. infusions once daily for 20 days followed by oral treatment 600 mg × 3 daily for 140 days.

ELIGIBILITY:
Inclusion Criteria:

The medical condition / disease to be studied is symptomatic diabetic peripheral polyneuropathy.

All inclusion criteria must be answered "yes" for a patient to participate in the trial.

1. Has the patient given informed consent according to local requirements before any trial related activities? A trial related activity is any procedure that would not have been performed during the routine management of the patient.
2. Is the patient aged ≥ 18 to ≤ 65 years?
3. Does the patient suffer from type 2 diabetes mellitus?
4. Has the patient evidence of symptomatic diabetic peripheral polyneuropathy, i.e. TSS ≥ 6 and NIS-LL ≥ 2?
5. Is the patient's VPT measured to ≤ 30V?
6. Has the patient adequate circulation to the foot as evidenced by a palpable pulse on posterior tibialis artery and dorsal artery of foot?
7. Is the HbA1C level less than 10%?
8. Is the patient able to make frequent clinic visits over the trial period?

   For patients receiving tricyclic antidepressants, anticonvulsants, mexiletine or neuroleptics as treatment of neuropathic pain:
9. Has the regimen been stable within the last month?

   For female patients of childbearing potential (childbearing potential is considered until menopause has lasted more than 12 months):
10. Does the patient use an acceptable contraceptive method (hormonal pills, patches, implants, injections or intrauterine device)?
11. Is the pregnancy test negative before the 1st dose of trial medication?

(Surgically hysterectomised and surgically successfully sterilized females may be included on the same conditions as male patients).

Exclusion Criteria:

All exclusion criteria must be answered "no" for a patient to participate in the trial.

1. Does the patient suffer from known allergy towards Actovegin or similar preparations?
2. Has the patient asymmetrical neuropathy of the trunk or proximal lower limbs?
3. Does the patient suffer from diabetic foot ulceration or infections?
4. Does the patient suffer from diabetic amyotrophy?
5. Does the patient suffer from decompensated cardiac insufficiency, pulmonary oedema, oliguria, anuria, generalised oedema?
6. Does the patient suffer from polyneuropathy due to other underlying causes?
7. Has the patient been hospitalised due to diabetic polyneuropathy within the last month?
8. Has the patient participated in any other trial with an Investigational Medicinal Product (IMP) or device within 30 days before inclusion in this trial?
9. Has the patient ever used medications that may be etiological factors for neuropathy, such as isoniazid, nitrofurantoin, vincristine and phenytoin?
10. Has the patient used cerebrolysin or α-lipoic acid or received Transcutaneous Electric Nerve Stimulation (TENS) or acupuncture within the last month?
11. Has the patient received opiates as treatment of his / her diabetic polyneuropathy within the last month?
12. Does the patient suffer from any malignancy?
13. Is the patient nursing?
14. Does the patient suffer from any mental, psychiatric or other conditions that may compromise data collection and understanding of written and verbal information given in the trial?
15. Does the patient suffer from present and / or previous chronic alcohol abuse?
16. Is there any anamnestic evidence of hypothyroidism?
17. Is there any anamnestic evidence of vitamin B12 deficiency?
18. Does the patient suffer from an impaired renal function with high blood urea nitrogen (BUN) and / or increased serum creatinine (>120 µmol/L)?

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
TSSaverage: Average of the TSS over the treatment period (AUC / exposure time) VPTaverage: Average of the VPT measurement over the treatment period (AUC / exposure time) | Approx. 5½ months

SECONDARY OUTCOMES:
NIS-LLaverage: Average of the NIS-LL over the treatment period (AUC / exposure time) | Approx. 5½ months

CONTACTS AND LOCATIONS:
Overall Officials: Nycomced Clinical Trial Operations, Study Chair — Headquaters
Locations (1):
- Nycomed, Roskilde, Denmark